CLINICAL TRIAL: NCT00487539
Title: A Phase 2/3 Multicenter, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Safety and Efficacy of Golimumab Induction Therapy, Administered Subcutaneously, in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: An Efficacy and Safety Study of Golimumab (CNTO 148) in Participants With Moderately to Severely Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR014176; C0524T17; 2006-003398-28 (EudraCT Number); NCT00487539 (Registry Identifier: ClinicalTrials.gov Identifier)
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Colitis, Ulcerative
Keywords: Colitis, Ulcerative; Golimumab; CNTO 148
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo subcutaneous injection (given under the skin by way of a needle) matching to golimumab administered at Week 0 and Week 2.
  Interventions: Biological: Placebo
- Golimumab 100 mg -> 50 mg (Experimental): Golimumab 100 milligram (mg) subcutaneous injection administered at Week 0 and dose is decreased to 50 mg at Week 2.
  Interventions: Biological: Golimumab 100 mg; Biological: Golimumab 50 mg
- Golimumab 200 mg -> 100 mg (Experimental): Golimumab 200 mg subcutaneous injection administered at Week 0 and dose is decreased to 100 mg at Week 2.
  Interventions: Biological: Golimumab 100 mg; Biological: Golimumab 200 mg
- Golimumab 400 mg -> 200 mg (Experimental): Golimumab 400 mg subcutaneous injection administered at Week 0 and dose is decreased to 200 mg at Week 2.
  Interventions: Biological: Golimumab 200 mg; Biological: Golimumab 400 mg

INTERVENTIONS:
Biological: Placebo — Placebo subcutaneous injection (given under the skin by way of a needle) matching to golimumab administered at Week 0 and Week 2.
  Arms: Placebo
Biological: Golimumab 100 mg — Golimumab 100 mg subcutaneous injection administered at Week 0 for Golimumab 100 mg -> 50 mg arm group and at Week 2 for Golimumab 200 mg -> 100 mg arm group.
  Arms: Golimumab 100 mg -> 50 mg; Golimumab 200 mg -> 100 mg
Biological: Golimumab 200 mg — Golimumab 200 mg subcutaneous injection administered at Week 0 for Golimumab 200 mg -> 100 mg arm group and at Week 2 for Golimumab 400 mg -> 200 mg arm group.
  Arms: Golimumab 200 mg -> 100 mg; Golimumab 400 mg -> 200 mg
Biological: Golimumab 400 mg — Golimumab 400 mg subcutaneous injection administered at Week 0 for Golimumab 400 mg -> 200 mg arm group.
  Arms: Golimumab 400 mg -> 200 mg
Biological: Golimumab 50 mg — Golimumab 50 mg subcutaneous injection administered at Week 2 for Golimumab 100 mg -> 50 mg arm group.
  Arms: Golimumab 100 mg -> 50 mg

SUMMARY:
The purpose of this study is to assess the effects (good and bad) of golimumab (CNTO 148) therapy in participants with ulcerative colitis (UC).

DETAILED DESCRIPTION:
This is a multi-center (conducted in more than one center), randomized (study medication assigned by chance), double-blind (neither the physician nor the participant know about the study medication), placebo-controlled (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), parallel-group (a medical research study comparing the response in 2 or more groups of participants receiving different interventions) study to evaluate the safety and efficacy of golimumab in participants with moderately to severely active UC. There are 2 parts in this study. Part 1 is "Phase 2 dose-ranging" portion of study. Participants enrolled in Part 1, will receive subcutaneous (under the skin by way of a needle) injections of placebo, golimumab 100 milligram (mg), 200 mg, or 400 mg at Week 0, followed by subcutaneous injections of placebo, golimumab 50 mg, 100 mg, or 200 mg respectively at Week 2. Part 2 is "Phase 3 dose-confirming" portion of study and newly enrolled participants will receive same doses studied in Part 1, until the doses for Part 2 are selected. At the time that the final doses are selected, all newly enrolled participants will receive 1 of the selected doses or matching placebo. At Week 6, participants will be asked to participate in an additional 1-year maintenance study. Participants not entering the 1-year golimumab maintenance study will be evaluated for safety 16 weeks after last administration of study agent. The duration of study will be 6 weeks for participants who enter the 1-year golimumab maintenance study and 16 weeks after last administration of study agent for participants who do not enter the 1-year golimumab maintenance study. Efficacy of the participants will primarily be evaluated by clinical response at Week 6. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with moderately to severely active ulcerative colitis (UC) defined by a Mayo score of 6 to 12 inclusive at Baseline (Week 0), including an endoscopic (examination of an internal part of the body with a lighted tube; looking at a part of the body with a lighted tube) subscore of greater than or equal to 2
* Participants must have biopsy results (collected at the screening endoscopy (procedure or obtained within the last year) consistent with the diagnosis of UC
* Participants either currently receiving treatment with, or have a history of failure to respond to, or tolerate, at least 1 of the following therapies: oral 5-aminosalicylate, oral corticosteroids, 6-mercaptopurine and azathioprine
* Participants with current dependency or with a history of corticosteroid dependency (i.e., an inability to successfully taper corticosteroids without a return of the symptoms of UC)
* Not have a diagnosis of active tuberculosis
* Participants with negative stool test for enteric (by way of the intestines) pathogens

Exclusion Criteria:

* Participants with prior exposure to biologic anti-tumor necrosis factor (TNF) agents
* Participants with severe extensive UC that is likely to require a colectomy (surgery to remove part or all of the colon) within 12 weeks of study entry
* Participants having UC limited to the rectum only or to less than 20 centimeter of the colon
* Presence of a stoma (an artificial permanent opening especially in the abdominal wall made in surgical procedures) or presence of a fistula
* Participants with a history of extensive colonic resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1065 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (200):
- United States (58):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Roseville, California
  - San Diego, California
  - Golden, Colorado
  - Newark, Delaware
  - Boca Raton, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - Port Orange, Florida
  - Winter Park, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Clive, Iowa
  - Pratt, Kansas
  - Lexington, Kentucky
  - Monroe, Louisiana
  - Ann Arbor, Michigan
  - Troy, Michigan
  - Rochester, Minnesota
  - Pascagoula, Mississippi
  - Tupelo, Mississippi
  - Egg Harbor, New Jersey
  - New York, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Morganton, North Carolina
  - New Bern, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Colombus, Ohio
  - Norman, Oklahoma
  - Portland, Oregon
  - Limerick, Pennsylvania
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Sugar Land, Texas
  - Logan, Utah
  - Ogden, Utah
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Richmond, Virginia
  - Spokane, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (8):
  - Bankstown
  - Box Hill
  - Fitzroy
  - Herston
  - Launceston
  - Parkville
  - Prahran
  - Westmead
- Vienna, Austria
- Belgium (5):
  - Brussels
  - Ghent
  - Leuven
  - Liège
  - Roeselare
- Bulgaria (3):
  - Pleven
  - Rousse
  - Sofia
- Canada (8):
  - Vancouver, British Columbia
  - Barrie, Ontario
  - Chatham, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Saskatoon, Saskatchewan
  - T2n
  - Windsor
- Czechia (4):
  - Èeské Budìjovice 1
  - Hradec Králové
  - Litoměřice
  - Ostrava
- Denmark (4):
  - Aalborg
  - Aarhus C
  - Hvidovre
  - Odense C
- France (5):
  - Amiens Cedex 1 80
  - Bordeaux
  - Lille
  - Nice
  - Paris
- Germany (11):
  - Berlin
  - Berlin Be
  - Bochum
  - Hamburg
  - Hanover
  - Haßloch
  - Kiel
  - Minden
  - München
  - Münster
  - Stade
- Hungary (11):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Dunaújváros
  - Gyulai Ut 18
  - Mosonmagyaróvár
  - Sopron
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Veszprém
- India (8):
  - Bangalore
  - Chennai
  - Hyderabad
  - Hyderabad Andh Prad
  - Kārnād
  - New Delhi
  - Pune
  - Vishakapatanam
- Israel (9):
  - Beer Yaakov
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Nazareth
  - Petah-Tikv
  - Rehovot
  - Tel Aviv
- Japan (15):
  - Bunkyō City
  - Chikushinoshi
  - Fukuoka
  - Hiroshima
  - Kagoshima
  - Kurashiki
  - Kurume
  - Nagoya
  - Nishinomiya
  - Okayama
  - Osaka
  - Sakura
  - Sapporo
  - Tokyo
  - Yokkaichi
- Lithuania (2):
  - Kaunas
  - Vilnius
- Netherlands (4):
  - Amsterdam
  - Ede Gld
  - Groningen
  - Leiden
- New Zealand (3):
  - Christchurch
  - Dunedin
  - Hamilton
- Poland (12):
  - Bydgoszcz
  - Częstochowa
  - Elblag
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Opole
  - Sopot
  - Szczecin
  - Torun
  - Warsaw
- Romania (5):
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Târgu Mureş
  - Timișoara
- Russia (5):
  - Moscow
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Yaroslavl
- Serbia (3):
  - Belgrade
  - Niš
  - Zemun
- Slovakia (5):
  - Bratislava
  - Martin
  - Nitra
  - Nové Mesto nad Váhom
  - Prešov
- South Africa (4):
  - Cape Town
  - Cape Town West Cape
  - Marianhill Kz-Natal
  - Pretoria Gauteng
- Stockholm, Sweden
- Ukraine (6):
  - Donetsk
  - Kharkiv
  - Kyiv
  - Simferopol
  - Vynnytsya
  - Zhaporozhia 69104

REFERENCES:
- [Derived] Adedokun OJ, Xu Z, Liao S, Strauss R, Reinisch W, Feagan BG, Sandborn WJ. Population Pharmacokinetics and Exposure-Response Modeling of Golimumab in Adults With Moderately to Severely Active Ulcerative Colitis. Clin Ther. 2020 Jan;42(1):157-174.e4. doi: 10.1016/j.clinthera.2019.11.010. Epub 2020 Jan 22. PMID 31982148
- [Derived] Li K, Strauss R, Marano C, Greenbaum LE, Friedman JR, Peyrin-Biroulet L, Brodmerkel C, De Hertogh G. A Simplified Definition of Histologic Improvement in Ulcerative Colitis and its Association With Disease Outcomes up to 30 Weeks from Initiation of Therapy: Post Hoc Analysis of Three Clinical Trials. J Crohns Colitis. 2019 Aug 14;13(8):1025-1035. doi: 10.1093/ecco-jcc/jjz022. PMID 30721964
- [Derived] Sandborn WJ, Feagan BG, Marano C, Zhang H, Strauss R, Johanns J, Adedokun OJ, Guzzo C, Colombel JF, Reinisch W, Gibson PR, Collins J, Jarnerot G, Hibi T, Rutgeerts P; PURSUIT-SC Study Group. Subcutaneous golimumab induces clinical response and remission in patients with moderate-to-severe ulcerative colitis. Gastroenterology. 2014 Jan;146(1):85-95; quiz e14-5. doi: 10.1053/j.gastro.2013.05.048. Epub 2013 Jun 2. PMID 23735746

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to Placebo, Golimumab 100 mg->50 mg, Golimumab 200 mg->100 mg and Golimumab 400 mg->200 mg groups for dose selection. Efficacy results were reported for only newly enrolled participants assigned to Placebo, Golimumab 200 mg->100 mg and Golimumab 400 mg->200 mg groups after dose-selection as per planned analysis.
Groups:
- Placebo: Placebo subcutaneous injection (given under the skin by way of a needle) matched to golimumab administered at Week 0 and Week 2. This dosing regimen was selected for the efficacy analysis (only in newly enrolled participants following dose-selection, as per planned analysis).
- Golimumab 100 mg -> 50 mg: Golimumab 100 milligram (mg) subcutaneous injection was administered at Week 0 and dose was decreased to 50 mg at Week 2.
- Golimumab 200 mg -> 100 mg: Golimumab 200 mg subcutaneous injection was administered at Week 0 and the dose was decreased to 100 mg at Week 2. This dosing regimen was selected for the efficacy analysis (only in newly enrolled participants following dose-selection, as per planned analysis).
- Golimumab 400 mg -> 200 mg: Golimumab 400 mg subcutaneous injection was administered at Week 0 and the dose was decreased to 200 mg at Week 2. This dosing regimen was selected for the efficacy analysis (only in newly enrolled participants following dose-selection, as per planned analysis).
Period: Overall Study
Arm/Group | Placebo | Golimumab 100 mg -> 50 mg | Golimumab 200 mg -> 100 mg | Golimumab 400 mg -> 200 mg
Started | 331 | 72 | 331 | 331
Completed | 324 | 69 | 328 | 327
Not Completed | 7 | 3 | 3 | 4
Not completed — Adverse Event | 3 | 2 | 1 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 0 | 0 | 1
Not completed — Other | 3 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo subcutaneous injection (given under the skin by way of a needle) matched to golimumab administered at Week 0 and Week 2.
- Golimumab 200 mg -> 100 mg: Golimumab 200 mg subcutaneous injection was administered at Week 0 and dose was decreased to 100 mg at Week 2.
- Golimumab 400 mg -> 200 mg: Golimumab 400 mg subcutaneous injection was administered at Week 0 and dose was decreased to 200 mg at Week 2.
- Total: Total of all reporting groups
Arm/Group | Placebo | Golimumab 100 mg -> 50 mg | Golimumab 200 mg -> 100 mg | Golimumab 400 mg -> 200 mg | Total
Number analyzed (Participants) | 331 | 72 | 331 | 331 | 1065
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39 (13.04) | 40.9 (12.19) | 40 (13.54) | 40.7 (13.75) | 40 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 32 | 151 | 130 | 469
  Male | 175 | 40 | 180 | 201 | 596

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response at Week 6
Description: Clinical response is defined as decrease from baseline in Mayo score by greater than or equal to 30 percent and greater than or equal to 3, with either a decrease from baseline in rectal bleeding sub-score of greater than or equal to 1 or a rectal bleeding sub-score of 0 or 1. The Mayo score is sum of 4 sub-scores (i.e., stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total Mayo score value ranges from 0 to 12.
Time Frame: Baseline, Week 6
Population: Efficacy analysis population included all the participants who were randomly assigned to the study after the dose selection.
Measure: Number; unit: Participants
Arm/Group | Placebo | Golimumab 200 mg -> 100 mg | Golimumab 400 mg -> 200 mg
Number analyzed (Participants) | 251 | 253 | 257
Participants | 76 | 129 | 141
Statistical Analysis 1: Comparison: Placebo vs Golimumab 200 mg -> 100 mg; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Golimumab 400 mg -> 200 mg; Test type: Superiority or Other; p < 0.0001, Chi-squared

2. Secondary Outcome: Number of Participants With Clinical Remission at Week 6
Description: Clinical remission is defined as a Mayo score of less than or equal to 2, with no individual sub-score greater than 1. The Mayo score is sum of 4 sub-scores (i.e., stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total Mayo score value ranges from 0 to 12.
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Golimumab 200 mg -> 100 mg | Golimumab 400 mg -> 200 mg
Number analyzed (Participants) | 251 | 253 | 257
Participants | 16 | 45 | 46
Statistical Analysis 1: Comparison: Placebo vs Golimumab 200 mg -> 100 mg; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Golimumab 400 mg -> 200 mg; Test type: Superiority or Other; p < 0.0001, Chi-squared

3. Secondary Outcome: Number of Participants With Mucosal Healing at Week 6
Description: Mucosal healing is determined from the endoscopy sub-score of the Mayo score. Mucosal healing is defined as an endoscopy sub-score of 0 or 1. Higher score indicates higher severity of disease. Endoscopy sub-score ranges from 0 (normal or inactive disease) to 3 (severe disease; spontaneous bleeding and ulceration).
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Golimumab 200 mg -> 100 mg | Golimumab 400 mg -> 200 mg
Number analyzed (Participants) | 251 | 253 | 257
Participants | 72 | 107 | 116
Statistical Analysis 1: Comparison: Placebo vs Golimumab 200 mg -> 100 mg; Test type: Superiority or Other; p = 0.0014, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Golimumab 400 mg -> 200 mg; Test type: Superiority or Other; p = 0.0001, Chi-squared

4. Secondary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 6
Description: The IBDQ is used to measure disease specific quality of life on a 32 Likert-scaled items questionnaire. The IBDQ scale contains 4 component subscales: bowel symptoms, systemic symptoms, emotional function and social function with scores ranging from 10 to 70, 5 to 35, 12 to 84 and 5 to 35 respectively and the total score ranges from 32 to 224. Higher scores indicate better health related quality of life.
Time Frame: Baseline to Week 6
Population: Efficacy analysis population included all the participants who were randomly assigned to the study after the dose selection. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Golimumab 200 mg -> 100 mg | Golimumab 400 mg -> 200 mg
Number analyzed (Participants) | 250 | 252 | 255
Units on a Scale
  Baseline | 129.6 (32.61) | 131.7 (33.93) | 127.2 (33.90)
  Change at Week 6 | 14.8 (31.25) | 27.0 (33.72) | 26.9 (34.28)
Statistical Analysis 1: Comparison: Placebo vs Golimumab 200 mg -> 100 mg; Test type: Superiority or Other; p < 0.0001, ANOVA; on the van der Waerden normal scores
Statistical Analysis 2: Comparison: Placebo vs Golimumab 400 mg -> 200 mg; Test type: Superiority or Other; p < 0.0001, ANOVA; on the van der Waerden normal scores

ADVERSE EVENTS:
Time Frame: 6 weeks for participants who entered the maintenance study. 16 weeks following the last study agent administration for participants who did not enter the maintenance study.
Description: The safety population reflects the "as treated" population: 1 participant out of the 331 randomized to placebo, received golimumab 100 mg at Week 0 and is included in the 200 mg -> 100 mg group; 1 participant out of the 331 randomized to the 200 mg -> 100 mg group, received 200 mg golimumab at Week 2 and is included in the 400 mg -> 200 mg group.
Arm/Group | Placebo | Golimumab 100 mg -> 50 mg | Golimumab 200 mg -> 100 mg | Golimumab 400 mg -> 200 mg
Serious Adverse Events (participants affected / at risk) | 20/330 | 3/71 | 10/331 | 15/332
Other Adverse Events (participants affected / at risk) | 61/330 | 18/71 | 54/331 | 55/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=330) | Golimumab 100 mg -> 50 mg (N=71) | Golimumab 200 mg -> 100 mg (N=331) | Golimumab 400 mg -> 200 mg (N=332)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 8 | 1 | 3 | 7
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Adverse Drug Reaction (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Anal Abscess (Infections and infestations) | 1 | 0 | 0 | 1
Brain Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Cytomegalovirus Infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1
Haematoma Infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes Simplex (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Rectal Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 1 | 0
Volume Blood Decreased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Carcinoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Demyelination (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=330) | Golimumab 100 mg -> 50 mg (N=71) | Golimumab 200 mg -> 100 mg (N=331) | Golimumab 400 mg -> 200 mg (N=332)
Anaemia (Blood and lymphatic system disorders) | 6 | 2 | 8 | 5
Abdominal Pain (Gastrointestinal disorders) | 5 | 1 | 2 | 7
Colitis Ulcerative (Gastrointestinal disorders) | 7 | 1 | 4 | 2
Nausea (Gastrointestinal disorders) | 6 | 1 | 3 | 12
Injection Site Erythema (General disorders) | 0 | 3 | 5 | 4
Pyrexia (General disorders) | 7 | 2 | 5 | 10
Nasopharyngitis (Infections and infestations) | 12 | 2 | 13 | 8
Oral Herpes (Infections and infestations) | 1 | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0 | 3 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1
Headache (Nervous system disorders) | 17 | 5 | 11 | 15
Insomnia (Psychiatric disorders) | 3 | 2 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
12 months after study ends, Sponsor will be provided with a copy of the materials at least 45 days prior to submission, with details of proposed date, journal or conference name of publication & it will have 30 days post receipt to send a written request that the publication be delayed on the basis it exposes intellectual property that requires propriety protection but it will be only for 60 days after which Investigator will be free to publish. The participation of Sponsor will be acknowledged.